CLINICAL TRIAL: NCT05520021
Title: Comparison of the Effects of Nifedipine and Magnesium Sulfate on Maternal and Fetal Doppler Blood Flow Patterns in Women With Preterm Labor
Brief Title: The Treatment of Magnesium Sulfate and Nifedipine in Preterm Labor Threat
Acronym: MgSO4
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Konya Meram State Hospital (Other)
Responsible Party: Principal Investigator, Hasan Ali Inal, MD, Clinical Professor, Konya Meram State Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 351507
Record Dates: First submitted 2022-08-25; First posted 2022-08-29 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-08

CONDITIONS: Preterm Labor Without Delivery; Pregnancy Preterm
Keywords: Nifedipine; Magnesium sulfate; pregnancy; preterm labor threat
MeSH Terms: interventions — Nifedipine; Magnesium Sulfate

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Magnesium sulfate treatment (Active Comparator): A total of 30 pregnancies with preterm labor threats will be treated with Magnesium sulfate.
  Interventions: Drug: Magnesium sulfate
- Nifedipine treatment (Active Comparator): A total of 30 pregnancies with preterm labor threats will be treated with Nifedipine.
  Interventions: Drug: Nifedipine
- Healthy pregnant women (No Intervention): A total of 30 pregnancies without preterm labor threat will be included.

INTERVENTIONS:
Drug: Nifedipine — A total of 30 pregnancies with preterm labor threats will be treated with Nifedipine.
  Arms: Nifedipine treatment
Drug: Magnesium sulfate — A total of 30 pregnancies with preterm labor threats will be treated with Magnesium sulfate.
  Arms: Magnesium sulfate treatment

SUMMARY:
Comparison of the effects of Nifedipine and MgSO4 therapies on maternal and fetal blood flow.

DETAILED DESCRIPTION:
In this study, the investigators aim to compare the effect of Nifedipine and MgSO4 therapies on Doppler parameters of the uterine, umbilical, middle cerebral arteries, and ductus venous in the first 48 hours of therapy in pregnancies with preterm labor threat and also compare perinatal outcomes after delivery between the groups.

ELIGIBILITY:
Inclusion Criteria:

* pregnancies with preterm labor threat between 28-34 weeks gestational ages

Exclusion Criteria:

* Cervical dilatation at > 4 cm and/or cervical effacement >80%,
* Multiple pregnancies,
* Pregnancy complications including preeclampsia, ablatio placenta, intrauterine growth restriction, placenta previa, gestational diabetes

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Doppler parameters | Gestational age at delivery (weeks)
  Pulsality index of middle cerebral artery.

SECONDARY OUTCOMES:
Perinatal outcomes | Gestational age at delivery (weeks)
  NICU admission

CONTACTS AND LOCATIONS:
Overall Officials: Hasan A Inal, Principal Investigator — Antalya Training and Research Hospital
Locations (1):
- Hasan Ali Inal, Antalya, Turkey (Türkiye)